CLINICAL TRIAL: NCT07282678
Title: Closed-Loop Transcranial Alternating Current Stimulation for the Treatment of Major Depressive Disorder: Double-Blind, Controlled Randomized Multicenter Clinical Trial
Brief Title: Closed-Loop Transcranial Alternating Current Stimulation for the Treatment of Major Depressive Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pulvinar Neuro, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PN1000
Record Dates: First submitted 2025-12-05; First posted 2025-12-15 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Depression - Major Depressive Disorder; Transcranial Alternating Current Stimulation
Keywords: tACS; Depression; Major Depressive Disorder; Transcranial Alternating Current Stimulation
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Active Closed-loop tACS (Experimental): Closed-loop individual alpha tACS daily for five consecutive days.
  Interventions: Device: Closed-loop tACS
- Sham Closed-loop tACS (Sham Comparator): Sham closed-loop individual alpha tACS daily for five consecutive days.
  Interventions: Device: Sham Comparator
- Open Label, Active Closed-loop tACS Retreatment (Experimental): An open label, second dose of Closed-loop individual alpha tACS daily for five consecutive days. Assignment to this arm occurs after participation in the closed label active or sham arms.
  Interventions: Device: Closed-loop tACS

INTERVENTIONS:
Device: Closed-loop tACS — Individual alpha tACS
  Arms: Active Closed-loop tACS; Open Label, Active Closed-loop tACS Retreatment
Device: Sham Comparator — Sham stimulation
  Arms: Sham Closed-loop tACS

SUMMARY:
The purpose of this research study is to investigate a closed-loop transcranial alternating current stimulation (tACS) device to evaluate its ability to reduce symptoms of major depressive disorder

DETAILED DESCRIPTION:
This study examines the efficacy of closed-loop transcranial alternating current stimulation (CL-tACS) for the treatment of major depressive disorder (MDD) in a double-blind, controlled parallel group multi-site clinical trial. 214 participants will be randomized into receiving 5 consecutive days of active or control CL-tACS (1:1 allocation) to achieve approximately 192 participants completing the primary endpoint at week 3, assuming a 10% lost to follow-up rate. Clinical assessments of depression and anxiety symptoms are performed at Screening, Baseline, Day 5, Follow-Up 1 (week 3), and Follow-Up 2 (week 5). Additional assessments of quality of life are included.

For subjects who are not considered responders at the Week 3 primary endpoint, there will be a phase 2 retreatment with active CL-tACS which will mirror the same 5-day protocol. Patients in this arm will complete additional data collection at Phase 2 baseline, Phase 2 Day 5, Phase 2 Follow-up 1 (phase 2 week 3), and phase 2 follow-up 2 (phase 2 week 5).

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 22 years of age;
2. with at least moderate symptom severity (HAM-D17 ≥ 17);
3. who are currently in a depressive episode;
4. who have used at least 1 antidepressant in the current or previous episode, but have not found adequate symptom relief or who were not able to tolerate medication side effects;
5. who, for 6 weeks prior to enrollment, are either;

   * not taking antidepressant medication, or:
   * are taking a stable psychiatric medication regimen with one or more stable antidepressant medication dose(s)
6. if currently engaged in depression-focused psychotherapy, have maintained stable frequency of therapy for at least 8 weeks prior to enrollment and agree to continue the same regimen throughout study participation;
7. are able and willing to comply with the protocol and follow up schedule and protocol, in the opinion of the investigator;
8. who understand English and are able to provide written informed consent;
9. who are currently under the care of a psychiatric clinician or a primary care physician for major depressive disorder, and who agree to promptly inform the study staff of any change of psychiatric or mental health providers during study participation;
10. who agree to allow any and all forms of communication between the investigators/study staff and their current or past (within 2 years) healthcare providers;
11. who agree to provide the names and verifiable contact information (email and mailing addresses, mobile and/or land-line phone numbers, as applicable) for at least two persons (≥ age 18) who reside within a 60-minute drive of their residence and whom the research staff are at liberty to contact, as they deem necessary, to ensure participant safety for the duration of study participation;

Exclusion Criteria:

1. Subjects with current / past six months use of an external stimulation device for MDD, including electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS), cranial electrotherapy stimulation (CES), transcranial direct current stimulation (tDCS), deep brain stimulation (DBS), or other brain or cranial nerve stimulation;
2. Subjects with (lifetime) history of failure to response to an adequate trial of ECT, TMS, or implanted vagus nerve stimulation;
3. Subjects who currently receive esketamine, ketamine, or psilocybin treatment
4. Subjects who are pregnant or of childbearing potential and not using adequate contraception, as determined by the investigator;
5. Subjects who are breastfeeding.
6. Subjects whose current depressive episode had onset within 6 months post-partum;
7. Presence of active skin disorder on the forehead that could be exacerbated by stimulation electrodes in the opinion of the investigator.
8. Subjects with clinical or historical features which, in the opinion of the investigator, make them an inappropriate candidate for participation in this trial;
9. Subjects whose current depressive episode has not responded to 3 or more adequate trials of FDA approved antidepressant medications;
10. Subjects with current suicidal ideation with plan or intent, or suicidal behavior or preparation in the past 3 months, as determined by CSSRS assessment or by the Investigator;
11. Subjects with a history of epilepsy or unexplained seizures, as determined by the Investigator;
12. Subjects with a diagnosis or clinical history suggestive of bipolar disorder, hypomania, mania, or psychosis, as determined by the Investigator.
13. Subjects currently participating, or intending to participate (during the next 3 months) in another study involving an investigational drug or device treatment that, in the opinion of the investigator, could impact symptoms of MDD or use of the investigational device;
14. Subjects with a history of intracranial surgery;
15. Subjects with implanted neurostimulators, nonremovable or implanted electrical devices or intracranial metal objects, with the exception of dental metal;
16. Subjects with cognitive impairment or memory disorders, which, in the opinion of the investigator, could impact their ability to comply with study requirements;
17. Subjects currently meeting diagnostic criteria for obsessive compulsive disorder;
18. Subjects who meet DSM-V criteria for moderate/severe alcohol use disorder or other substance use disorders (except tobacco/nicotine) within the past 6 months as confirmed by the DIAMOND interview;
19. Subjects who meet DSM-V criteria for moderate/severe cannabis use disorder (CUD) within the past 6 months as confirmed by the DIAMOND interview. Subjects with recreational or prescription use (including medical marijuana cards) not considered moderate to severe CUD will be included.
20. Subjects with a current neurological condition or disease which, in the opinion of the investigator, is likely to manifest a depressive syndrome or symptoms that would substantially confound the diagnosis or serial assessment of major depressive disorder.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS) score reduction, Phase 1 Evaluation | Timeframe: Baseline to Week 3
  Response rates (at least 50% reduction in HDRS-D17 score) (0-52 score range, higher score is worse)

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS) Score reduction, at study end | At the phase 1, week 3 assessment OR at the phase 2, week 3 assessment.
  Response rates (at least 50% reduction in HDRS-17 score) for patients at their study completion. This will be evaluated by determining the percentage of patients from the active stimulation arm who can be classified as responders either at the phase 1, week 3 assessment OR at the phase 2, week 3 assessment. (0-52 score range, higher score is worse)
The State-Trait Anxiety Inventory (STAI) Score | Timeframe: Baseline to week 3, Phase 1
  Change in self-reported anxiety symptoms STAI Trait (score range is 20-80, higher is worse)
Hamilton Depression Rating Scale (HDRS) Remission Rate | Timeframe: Baseline to Week 3, Phase 1
  Remission rates (HDRS-17 score ≤ 7) (0-52 score range, higher score is worse)
Hamilton Depression Rating Scale (HDRS) Remission Rate at Baseline Evaluation | Timeframe: Baseline to Day 5
  Remission rates (HDRS-17 score ≤ 7) (0-52 score range, higher score is worse)
Responder rates (at least 50% reduction in Hamilton Depression Rating Scale (HDRS) score) | Timeframe: Baseline to Day 5
  Responder rates (at least 50% reduction in HDRS-17 score) (0-52 score range, higher score is worse)
Change in Hamilton Depression Rating Scale (HDRS) Score | Timeframe: Baseline to Day 5
  Change in HDRS-17 Score (0-52 score range, higher score is worse)
Change in mean Hamilton Depression Rating Scale (HDRS) Score | Timeframe: Baseline to Week 3
  Change in mean HDRS-17 Score (0-52 score range, higher score is worse)
Remission rates (Hamilton Depression Rating Scale (HDRS) score ≤ 7) | Timeframe: Baseline to Week 5
  Remission rates (HDRS-17 score ≤ 7) (0-52 score range, higher score is worse)
Responder rates (at least 50% reduction in Hamilton Depression Rating Scale (HDRS) score) | [Timeframe: Baseline to Week 5].
  Responder rates (at least 50% reduction in HDRS-17 score) (0-52 score range, higher score is worse)
Change in Hamilton Depression Rating Scale (HDRS) score | Timeframe: Baseline to Week 5
  Change in HDRS-17 (0-52 score range, higher score is worse)

CONTACTS AND LOCATIONS:
Overall Officials: Mark George, MD, Principal Investigator — Medical University of South Carolina

IPD SHARING:
Plan to Share IPD: No